CLINICAL TRIAL: NCT01510080
Title: Live Supervision Put to Test - Studies of Acceptance and Efficacy of Computer-assisted Live Supervision
Brief Title: Acceptance and Efficacy of Live Supervision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, Florian Weck, Principal Investigator, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WECK-012
Record Dates: First submitted 2011-12-12; First posted 2012-01-13 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Mental Disorders
Keywords: Computer-assisted live supervision; "Bug-in-the-eye" supervision; Delayed video-based supervision; Cognitive behavioral therapy supervision
MeSH Terms: conditions — Mental Disorders | interventions — Dental Occlusion; Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-assisted live supervision (Experimental): Supervisees assigned to this group will receive 8 sessions of computer-assisted live supervision and 4 sessions of delayed video-based supervision while treating 2 patients during 26 therapy sessions each. Computer-assisted live supervision is also known as "bug-in-the-eye" (BITE) supervision. The supervisor observes the therapy session with the help of a webcam and types messages on his computer. The instructions to the supervisee appear on a second monitor located in the therapy room where the supervisee can view it whenever he wants to.
  Interventions: Behavioral: Computer-assisted live supervision
- Delayed video-based supervision (Experimental): Supervisees assigned to this group will receive 12 sessions of delayed video-based supervision while treating 2 patients during 26 therapy sessions each. During delayed video-based supervision the supervisor and the supervisee spend 50 minutes reviewing selected parts of video recorded therapy sessions and discussing the case.
  Interventions: Behavioral: Delayed video-based supervision

INTERVENTIONS:
Behavioral: Computer-assisted live supervision — 8 BITE sessions, 4 video-based sessions (each 50 minutes) during treatment of 2 patients
  Other Names: "bug-in-the-eye" (BITE) supervision; video-based live supervision; monitor-based live supervision
  Arms: Computer-assisted live supervision
Behavioral: Delayed video-based supervision — 12 video-based sessions (each 50 minutes) during treatment of 2 patients
  Other Names: videotape supervision
  Arms: Delayed video-based supervision

SUMMARY:
In order to meet an existing lack of empirical studies in the field of cognitive behavioral therapy supervision, the present randomized controlled trial is aimed at comparing two different types of supervision. This study compares computer-assisted live supervision and delayed video-based supervision regarding efficacy and acceptance among therapists, patients and supervisors. The efficacy of supervision is defined on different levels such as change of psychotherapeutic competence, nondisclosure, self-efficacy, self-awareness of the supervisee as well as therapeutic alliance, supervisory alliance and therapy outcome.

ELIGIBILITY:
Supervisees

Inclusion Criteria:

* Having successfully completed the interim audit
* Having started to treat ambulant patients under supervision

Exclusion Criteria:

-

Patients

Inclusion Criteria:

* Meeting ICD 10 criteria for a mental disorder
* Informed consent

Exclusion Criteria:

* Currently in psychotherapy
* Suicidal tendency
* Clinical diagnosis of alcohol or drug addiction, acute schizophrenia, schizoaffective disorder or bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Supervisory Questionnaire (SQ) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses nondisclosure of the supervisee during supervision
Supervisee Levels Questionnaire (SLQ-R) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses self awareness, motivation and dependency- autonomy of supervisees
Counseling Self-Estimate Inventory (COSE) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses self efficacy of the supervisee
Fragebogen zur Psychotherapie-Supervision Kurzform (FSPT-K) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses level of development and supervision needs of the therapist

SECONDARY OUTCOMES:
Helping Alliance Questionnaire (HAQ) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses the therapeutic alliance
Supervisory Working Alliance Inventory (SWAI) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses the supervisory relationship
Beck-Depression Inventory II (BDI-II) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses depressive symptoms
Beck Anxiety Inventory II (BAI) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that asessses anxiety symptoms
Brief Symptom Inventory (BSI) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses aspects of general psychopathology
Health-related quality of life (SF-12) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses the health-related quality of life
Client Satisfaction Questionnaire (CSQ8) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses satisfaction with therapy
Stundenbogen zur Supervisionsbeurteilung (STEP SV) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  self-report measure that assesses satisfaction with supervision
Cognitive Therapy Scale (CTS) | participants will be followed for the duration of psychotherapy, an expected average of 30 weeks
  clinician-rated measure that assesses psychotherapeutic competencies

CONTACTS AND LOCATIONS:
Overall Officials: Florian Weck, PhD, Principal Investigator — Goethe University; Martin Bohus, MD, Study Director — Central Institute of Mental Health
Locations (1):
- Department of Clinical Psychology and Psychotherapy of the Wolfgang Goethe University, Frankfurt am Main, Hesse, Germany